CLINICAL TRIAL: NCT06643117
Title: A Multicenter, Randomized, Double-blind Trial to Demonstrate Similar Efficacy, Safety, and Immunogenicity of FYB206 (Keytruda Biosimilar Candidate) in Comparison to Keytruda (Pembrolizumab) as an Add-on to Chemotherapy in Treatment-naïve Patients With Metastatic Non-squamous Non-small Cell Lung Cancer
Brief Title: Similar Efficacy, Safety, and Immunogenicity of FYB206 in Comparison to Keytruda as add-on to Chemotherapy in Patients With Non-squamous Non-small Cell Lung Cancer (NSCLC)
Acronym: Lotus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Formycon concluded that continuing the trial is no longer necessary for the development and approval of FYB206. The therapeutic comparability of FYB206 to Keytruda can be demonstrated based on comprehensive analytical and PK comparability data
Sponsor: Formycon AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FYB206-C3-02; 2023-509766-37-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-13; First posted 2024-10-16 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Non Small Cell Lung Cancer; Non-Squamous Non-Small Cell Lung Cancer
Keywords: pembrolizumab; biosimilar; lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- FYB206 (Experimental)
  Interventions: Biological: FYB206
- Keytruda (Active Comparator)
  Interventions: Biological: Keytruda

INTERVENTIONS:
Biological: FYB206 — FYB206 (Keytruda biosimilar candidate - test product) 200 mg administered as an IV infusion over 30 minutes on Day 1 of each cycle combined with chemotherapy in the first year (treatment Cycles 1 to 17)
  Arms: FYB206
Biological: FYB206 — Open-label treatment with FYB206 combined with chemotherapy (Cycles 18-34) to assure treatment continuation for trial patients up to a total of 2 years (a total of 34 treatment cycles)
  Arms: FYB206
Biological: Keytruda — Keytruda (reference product) 200 mg administered as an IV infusion over 30 minutes on Day 1 of each cycle combined with chemotherapy in the first year (treatment Cycles 1 to 17)
  Arms: Keytruda

SUMMARY:
NSCLC is the most common type of lung cancer. Metastatic cancers are cancers that start to spread to other parts of the body. NSCLC is treated by radiation therapy, with medicines, surgery, or immunotherapy. Immunotherapy is a type of treatment that helps the immune system fight cancer.

The immune system helps the body fight infections and disease. Pembrolizumab is an anti-cancer therapy that works with the immune system to fight cancer cells. Some cancer cells develop a way to hide from the body's immune system and, thus, allow the cancer cells to spread and grow. Pembrolizumab helps the immune system recognize and kill these cancer cells that want to hide. Pembrolizumab is a biologic drug (produced by living organisms) available in the market under the brand name Keytruda. Keytruda is approved globally for the treatment of a variety of cancers and as an addon or after therapy to primary cancer treatment like surgery. This helps prevent the cancer from returning, improving overall survival.

FYB206 is a proposed biosimilar to Keytruda. A biosimilar is not identical, but very similar to its original biologic. Biosimilars are expected to have a similar effect and safety to the original biologic. This clinical trial is intended to demonstrate the comparable effectiveness and safety of FYB206 to Keytruda as an add-on treatment to chemotherapy in patients with metastatic NSCLC who have not received previous anti-cancer treatment that is given directly into the blood.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed or cytologically confirmed diagnosis of Stage IV non-squamous NSCLC.
* Confirmation that epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK)-directed therapy is not indicated (ie, documentation of absence of tumor-activating/sensitizing EGFR mutations AND absence of ALK gene rearrangements).
* No prior systemic treatment for metastatic non-squamous NSCLC. Patients who received adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 12 months prior to the development of metastatic disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Small cell lung cancer (SCLC) or combination of SCLC and NSCLC. Squamous cell tumors and mixed adenosquamous carcinomas of predominantly squamous nature.
* Known one of the mutations listed below:

  * ROS1 fusion gene
  * BRAF-V600E
  * RET fusion
  * MET Exon 14
* Known active central nervous system metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are clinically stable for at least 2 weeks and have no evidence of new or enlarging brain metastases and are also off steroids 3 days prior to dosing with trial treatment. Stable brain metastases by this definition should be established prior to the first dose of trial treatment. Patients with known untreated, asymptomatic brain metastases (ie, no neurological symptoms, no requirements for corticosteroids, no or minimal surrounding edema, and no lesion >1.5 cm) may participate but will require regular imaging of the brain as a site of disease.
* Prior treatment with any anti-programmed cell death 1, PD-L1, or programmed cell death ligand 2 agent or an antibody targeting other immuno-regulatory receptors or mechanisms. Examples of such antibodies include (but are not limited to) antibodies against indoleamine 2, 3-dioxygenase, PD-L1, interleukin 2 receptor, or glucocorticoid-induced tumor necrosis factor receptor-related protein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Best objective response rate | 40 Weeks
  Best objective response rate (bORR): proportion of patients who had a best response of complete response (CR) or partial response (PR) as assessed by blinded independent central review (BICR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1

CONTACTS AND LOCATIONS:
Locations (13):
- Georgia (3):
  - Formycon Investigative Site, Batumi
  - Formycon Investigative Site, Kutaisi
  - Formycon Investigative Site, Tbilisi
- Malaysia (5):
  - Formycon Investigative Site, George Town
  - Formycon Investigative Site, Kuala Lumpur
  - Formycon Investigative Site, Kuching
  - Formycon Investigative Site, Shah Alam
  - Formycon Investigative Site, Subang Jaya
- Turkey (Türkiye) (5):
  - Formycon Investigative Site, Adana
  - Formycon Investigative Site, Diyarbakır
  - Formycon Investigative Site, Istanbul
  - Formycon Investigative Site, Izmir
  - Formycon Investigative Site, Samsun

IPD SHARING:
Plan to Share IPD: No